CLINICAL TRIAL: NCT05185674
Title: Sociodemographic,Clinical,Quality of Life, and Health Care Conditions After Hospital Discharge in Patients Who Required Admission to ICU for COVID-19 at Hospital Universitario Nacional Between April 2020 and March 2021. Bogotá, Colombia
Brief Title: Sociodemographic, Clinical, Quality of Life and Health Care Conditions in COVID-19 Survivors.
Status: Completed | Type: Observational
Sponsor: Javier Eslava (Other)
Responsible Party: Sponsor-Investigator, Javier Eslava, Principal Investigator. Professor, Universidad Nacional de Colombia
Organization: Universidad Nacional de Colombia (Other)
Other Study IDs: 53543 (Hermes); CEI-2021-06-01 (Other: Hospital Universitario Nacional de Colombia)
Record Dates: First submitted 2022-01-07; First posted 2022-01-11 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Post-acute COVID-19 Syndrome; Long-COVID; COVID-19; Long COVID; Post-acute Sequelae of SARS-CoV-2 Infection
Keywords: Sequelae; Quality of Life; Delivery of Health Care; Socioeconomic factors; Mental health; Functional status; Intensive Care Unit; COVID-19; Post-acute COVID-19 syndrome; Long-COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 survivors subjects: All patients discharged from the National University Hospital of Colombia (Bogotá, Colombia) who required admission to the Intensive Care Unit of the same institution with a confirmed diagnosis of SARS-CoV-2 disease (COVID-19 disease) between April 1, 2020 and March 31, 2021
  * Severe Acute Respiratory Syndrome (SARS)
  * Coronavirus (CoV)
  Interventions: Other: Exposure: Coronavirus disease 2019 (COVID-19)

INTERVENTIONS:
Other: Exposure: Coronavirus disease 2019 (COVID-19) — Having presented Coronavirus disease 2019 (COVID-19) and stay in the Intensive Care Unit

SUMMARY:
Sociodemographic, Clinical, Quality of Life, and Health Care Conditions After Hospital Discharge in Patients Who Required Admission to the Intensive Care Unit for COVID-19 at the Hospital Universitario Nacional Between April 2020 and March 2021. Bogotá, Colombia

The main objective of this study is to characterize the sociodemographic, clinical, quality of life and health care conditions in a cohort of patients who have survived a stay in the Intensive Care Unit of the National University Hospital of Colombia. Secondarily, associations between these findings and sociodemographic and clinical characteristics will be evaluated.

It is expected to contribute to the scientific literature through the characterization and epidemiology of the problem in a sample of patients from a Latin American country. It is planned to contribute not only with clinical data, but also with data on socioeconomic impacts on patients and notions of the health care they are receiving. Through the analyzes to be carried out, associations that will contribute to the evidence for prevention and management of the outcome will be explored.

DETAILED DESCRIPTION:
Progressively, the evidence is growing that COVID-19 survivors present persistent or new symptoms and / or alterations in diagnostic studies / functional tests. There is no consensual characterization and denomination for this outcome, proposing names such as "Long-COVID" or "Post-COVID Syndrome", among others. Nor are there homogeneous estimates regarding incidence and prevalence. Most of the population studies and surveys have been conducted in the United States, China, and European countries. It is considered that this problem can have negative effects on the quality of life, the health of patients and a significant burden of disease for the system. Patients may face inequities and barriers in health care.

At the national and global level; it is projected that large numbers of people may present or are exhibiting this "syndrome." Knowing the situation is necessary to formulate and develop responses in terms of prevention, diagnosis, management and rehabilitation.

This study will be carried out with the main purpose of characterizing the sociodemographic, clinical, quality of life and health care conditions in a cohort of patients who have survived a stay in the Intensive Care Unit of the National University Hospital of Colombia. Secondarily, associations between these findings and sociodemographic and clinical characteristics will be evaluated.

The study will be developed with patients who have been admitted to the Intensive Care Unit of the National University Hospital of Colombia for COVID-19. Once the study is explained to the potential participants, doubts are resolved and informed consent is obtained; clinical variables registered in the database will be taken and a remote interview (virtual, telephone) will be carried out with the participant applying the collection instrument that contains questions of own elaboration and validated and recognized scales. No physical, treatment or experimentation interventions will be made. The study period is from April 1, 2020 to March 31, 2021. A pilot test is included to determine the applicability of the collection instrument, average duration of the interview, feasibility of filling out informed consent by electronic means and disposition of the participants to receive the information and be part of the study.

The data is recorded in REDCap and will be taken to the R-Studio statistical program, through which and with the STATA v16.1 program the analysis will be executed.

As a benefit to patients, a copy of their answers to the instrument's medical questions and a medical guidance will be sent to them. It will be explained to the participants that said orientation does not replace a formal medical consultation nor does it correspond to a teleconsultation and medical orders will not be issued.

This study also corresponds to a Master's thesis in Public Health for the Universidad Nacional de Colombia, within the framework of the "Equidad en Salud" Research Group of the Universidad Nacional de Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria
* Living patients, who presented COVID-19 with admission to the Intensive Care Unit of the National University Hospital of Colombia between April 1, 2020 and March 31, 2021.
* Patients 18 years of age and older
* COVID-19 confirmed by polymerase chain reaction (PCR) test positive for SARS-CoV-19.
* Signature of informed consent

Exclusion Criteria:

* Missing data in the database, referring to the variables of interest
* Pregnant patients
* Limitation for communication in Spanish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: : Patients admitted to the Intensive Care Unit of the Hospital Universitario Nacional de Colombia (Bogotá, Colombia) between April 1, 2020 and March 31, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with new or persistent symptoms after COVID-19 Number of participants with new or persistent symptoms after COVID-19 | Baseline (At the time of the interview and application of the collection instrument)
  Percentage of Participants with one or more new or persistent symptoms. Assessment of the presence or absence of one or more new or persistent symptoms after having COVID-19, reported as yes or no for each symptom.
  If the participant manifests dyspnea, the severity will be evaluated using the Modified Medical Research Council (mMRC) instrument, with scoring options from 0 to 4. The higher score the worse the symptoms.
Health-related quality of life before and after presenting COVID-19 | Baseline (At the time of the interview and application of the collection instrument)
  The instrument 12-Item Short-Form Health Survey (SF-12v2) version in Spanish for Colombia will be applied. The valid questionnaire consists of 12 questions about mental and physical health. Questions will be asked for the current moment and also directed to before having COVID-19. Scores ranging from 0 to 100 with higher score indicating better health.
Health care conditions after presenting COVID-19 | Baseline (At the time of the interview and application of the collection instrument)
  The participants will be asked questions designed by the researchers in the collection instrument about medical controls that they have received after medical discharge from COVID-19 and mainly for new or persistent symptoms, reported as yes or no medical control. Frequency of each barrier in access to health services (by default in the collection instrument elaborated by researchers).
Socioeconomic impact after presenting COVID-19 | Baseline (At the time of the interview and application of the collection instrument)
  Frequency of each economic impact like salary decrease or job loss. The participants will be asked questions designed by the researchers in the collection instrument about possible personal socioeconomic impacts of having fallen ill with COVID-19 and being admitted to the Intensive Care Unit.
Mental health symptoms before and after presenting COVID-19 | Baseline (At the time of the interview and application of the collection instrument)
  The researchers use the valid instrument Self-Reporting Questionnaire (SRQ-20) version in Spanish. The scale consists of 20 questions to be answered: yes or no. The score ranges from 0-20, each positive answer add 1 point. Higher score indicating greater possibility of psychological distress.
Functional Independence before and after presenting COVID-19 | Baseline (At the time of the interview and application of the collection instrument)
  The Barthel Index, Spanish version, will be applied to assessment functional independence. Scores ranges from 0 to 100, when 100 is better outcome (independence) and 0 is worst outcome (total dependence).

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Loaiza-Fernandez, MD,MSc (c), Principal Investigator — Universidad Nacional de Colombia; Jairo A Pérez-Cely, MD, ICU, Principal Investigator — Hospital Universitario Nacional de Colombia / Universidad Nacional de Colombia; Javier H Eslava-Schamalbach, MD, PhD, Principal Investigator — Universidad Nacional de Colombia / Hospital Universitario Nacional de Colombia
Locations (1):
- Hospital Universitario Nacional de Colombia, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
Individual participant data are protected by legislation and by ethical standards for research.